CLINICAL TRIAL: NCT01591577
Title: Phase II Trial of Pulse Dosing of Lapatinib in Combination With Temozolomide and Regional Radiation Therapy for Upfront Treatment of Patients With Newly-Diagnosed Glioblastoma Multiforme
Brief Title: Lapatinib With Temozolomide and Regional Radiation Therapy for Patients With Newly-Diagnosed Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: GlaxoSmithKline (Industry); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-000493
Record Dates: First submitted 2012-05-02; First posted 2012-05-04 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Newly Diagnosed Glioblastoma Multiforme
MeSH Terms: interventions — Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lapatinib/Temozolomide/radiation (Experimental): Patients will be treated with a pulse dose of lapatinib every week and temozolomide 75 mg/m2 daily during radiation. Lapatinib will be administered beginning on the first day of radiation and temozolomide (+/-2 days). External beam fractionated regional radiation will be given on consecutive week days at 200 cGy daily doses to a total dose of 6000 cGy. Patients will have rest from temozolomide only for 2-4 weeks. Patients will continue with weekly pulse-dosing of lapatinib. After a 2-4 weeks rest(for temozolomide only) following completion of radiation therapy, temozolomide will be restarted as Cycle 1 at 150 mg/m2/day for 5 days out of every 28.Subsequent cycles can increase to 200 mg/m2/day as tolerated per investigator's judgment. Lapatinib pulse doses will be continued every week without interruption.Treatment will continue for 24 additional 28-day cycles of temozolomide if there is no evidence of progression.
  Interventions: Other: Lapatinib/Temozolomide/radiation

INTERVENTIONS:
Other: Lapatinib/Temozolomide/radiation — Patients will be treated with a pulse dose of lapatinib every week and temozolomide 75 mg/m2 daily during radiation. Lapatinib will be administered beginning on the first day of radiation and temozolomide (+/-2 days). External beam fractionated regional radiation will be given on consecutive week days at 200 cGy daily doses to a total dose of 6000 cGy. Patients will have rest from temozolomide only for 2-4 weeks. Patients will continue with weekly pulse-dosing of lapatinib. After a 2-4 weeks rest(for temozolomide only) following completion of radiation therapy, temozolomide will be restarted as Cycle 1 at 150 mg/m2/day for 5 days out of every 28.Subsequent cycles can increase to 200 mg/m2/day as tolerated per investigator's judgment. Lapatinib pulse doses will be continued every week without interruption.Treatment will continue for 24 additional 28-day cycles of temozolomide if there is no evidence of progression.

SUMMARY:
The purpose of this study is to test the safety and effects of a combination of a study drug, Lapatinib, plus the administration of standard radiation therapy and an FDA approved drug Temozolomide (chemotherapy agent) in patients with newly diagnozed glioblastoma Multiforme.Currently, only radiation therapy and Temozolomide chemotherapy are standard treatment for brain cancer.Lapatinib has not been FDA approved for use in brain tumors treatment. It has been approved to be used as a daily treatment with other chemotherapies by the FDA for the treatment of advanced breast cancer.

The purpose of this study is to find the answers to the following research questions:

1. Is Lapatinib given twice a week at higher dosages, with radiation therapy and Temozolomide, safe when given to patients with brain tumor?
2. What are the side effects of Lapatinib given twice a week at higher dosages when given with radiation therapy and Temozolomide and how often do they occur?
3. Can Lapatinib, radiation, and Temozolomide be effective in shrinking tumors when given to patients with brain tumors?
4. To determine whether the presence of genetic alterations specific proteins in the tumor samples can predict whether this study drug is effective on the tumor.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included in the study based on the following criteria:
* Patients will have histologically proven intracranial Glioblastoma Multiforme (GBM) or gliosarcoma (GS). This includes treatment-naïve patients with prior tissue diagnoses of lower grade gliomas that have been upgraded to GBM after repeat resection.
* Patients must have available archived tissues of 20-30 unstained slides. If frozen tissues are available, at least 200mg would be preferred, but not mandatory for study eligibility.
* Use of effective means of contraception (men and women) in subjects of child-bearing potential
* Cranial MRI or contrast CT must have been performed within 21 days of study entry. The use of MRI rather than CT is preferred. The same type of scan, i.e., MRI or CT must be used throughout the period of protocol treatment for tumor measurement. If the surgical procedure was a resection, cranial MRI or contrast CT performed within 96 hours of resection is preferred but not required. If the surgical procedure was a biopsy only, a head CT within 96 hours of the biopsy is acceptable. Patients without measurable or assessable disease are eligible.
* Patients must begin partial brain radiotherapy and temozolomide chemotherapy no sooner than 2 weeks and no later than 5 weeks from the surgery in which tissue was collected. Patients with GBM diagnosis from surgeries in which tissue was not collected will be eligible after repeat surgery performed to collect tissue, as long as no treatment has been initiated prior to surgery in which tissue was collected. In this case, initiation of treatment must begin within 2 to 5 weeks from the last surgery. Patients may have radiotherapy administered at outside facilities according to the specified guidelines (Appendix F). Radiotherapy must be given within 2 days of lapatinib initiation and by external beam to a partial brain field in daily fractions of 2.0 Gy, to a planned total dose to the tumor of 60.0 Gy in accordance with Appendix F. Stereotactic radiosurgery and brachytherapy will not be allowed.
* Patients must be willing to forego other drug therapy against the tumor while being treated with pulse dosing of lapatinib and temozolomide and radiation and subsequently pulse dosing lapatinib and temozolomide.
* All patients must sign an informed consent approved by the Institutional Review Board indicating that they are aware of the investigational nature of this study. Patients must sign an authorization for the release of their protected health information.
* Patients must be > 18 years old, and with a life expectancy > 12 weeks.
* Patients must have a Karnofsky performance status of > 60.
* Patients must have adequate bone marrow function (WBC > 3,000/µl, ANC > 1,500/mm3, platelet count of > 100,000/mm3, and hemoglobin > 10 gm/dl) and the test must be performed within 14 days prior to treatment initiation. Eligibility level for hemoglobin may be reached by transfusion.
* Patients must have adequate liver function (AST, ALT < 2.5 times ULN, and bilirubin < 1.5 times ULN) and the test must be performed within 14 days prior to treatment initiation.
* Patients must have adequate renal function (creatinine < 1.5 mg/dL) before starting therapy and the test must be performed within 14 days prior to treatment initiation.

EXCLUSION CRITERIA

* Patients who received previous radiotherapy to the brain.
* Patients who received cytotoxic drug therapy, non-cytotoxic drug therapy, or experimental drug therapy directed against the brain tumor. Patients who received Gliadel wafers will be excluded. Patients may have received or be receiving corticosteroids, analgesics, and other drugs to treat symptoms or prevent complications.
* Patients who may be receiving any EIAED (see Appendix C) within 2 weeks prior to registration, or any other prohibited medications within the Washout Period per Appendix D prior to registration. See section 6.5 for seizure medication managements.
* Patients with any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy.
* Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years are ineligible.
* Women who are pregnant (determined by high titer of serum beta-HCG) or Breast-feeding. (Women with reproductive potential must practice adequate contraception.)
* Patients who have any disease that will obscure toxicity or dangerously alter drug metabolism.
* Patients who have serious uncontrolled inter-current medical illness including, but not limited to, ongoing or active infection requiring IV antibiotics and psychiatric illness/social situations that would limit compliance with study requirements, or disorders associated with significant immunocompromised state (HIV, SLE, etc.).
* Patients who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-12-07 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2 years
  The primary objective is to estimate the overall survival in subjects with newly-diagnosed glioblastoma treated with lapatinib/temozolomide/radiation followed by lapatinib/temozolomide for 2 years or until progression is detected. If no progression is seen at 2 years, then single-agent lapatinib will be continued until progression.

CONTACTS AND LOCATIONS:
Overall Officials: Pioanh Nghiemphu, M D, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States

REFERENCES:
- [Derived] Yu A, Faiq N, Green S, Lai A, Green R, Hu J, Cloughesy TF, Mellinghoff I, Nghiemphu PL. Report of safety of pulse dosing of lapatinib with temozolomide and radiation therapy for newly-diagnosed glioblastoma in a pilot phase II study. J Neurooncol. 2017 Sep;134(2):357-362. doi: 10.1007/s11060-017-2533-6. Epub 2017 Jul 1. PMID 28669012